CLINICAL TRIAL: NCT02336724
Title: A Single Arm, Open Label, Multicenter, Phase II Study of Famitinib in Patients With Gastrointestinal Stromal Tumor
Brief Title: A Study of Famitinib in Patients With Gastrointestinal Stromal Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-II-GIST
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2016-01

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor; famitinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Famitinib (Experimental): 25 mg qd p.o.,28 days as one cycle,treatment discontinued when disease progression determined or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Famitinib

INTERVENTIONS:
Drug: Famitinib

SUMMARY:
Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study has shown that the toxicity is manageable.

The purpose of this study is to evaluate the efficacy and safety profile of Famitinib in patients with advanced or metastatic gastrointestinal stromal tumor who failed from imatinib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable advanced or metastatic, histologically-confirmed, gastrointestinal stromal tumor.Patients has been failed from last imatinib treatment due to disease progression or unacceptable toxicity and unable to use sunitinib.
* At least 2 weeks since the last imatinib administration
* Must have at least one measurable disease by RECIST1.1 criteria(tumour lesions ≥10mm in longest diameter, malignant lymph nodes ≥15mm in short axis, scanning layer ≤ 5 mm).
* ECOG Performance status 0-1
* Participants have adequate organ and marrow function as defined below:

neutrophils ≥ 1.5×10^9/L, platelets≥ 80×10^9/L, hemoglobin≥ 90g/L （no blood transfusion within 14 days), serum transaminase(ALT and AST ) ≤ 2.5×ULN (If liver metastases are present, serum transaminase≤5×ULN), total bilirubin ≤ 1.25×ULN, cholesterol ≤ 7.75mmol/L and triglyceride≤1 x ULN, creatinine ≤1x ULN,creatinine clearance rate > 50ml/min Urine protein ≥ + + and confirmed the 24-hour urinary protein>1.0 g normal serum calcium, potassium,magnesium, phosphorus INR≤1.5 and APTT≤1.5 ULN LVEF: ≥ 50%

* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy with tyrosine kinase -inhibitor agent targeting at VEGFR, PDGFR and c-Kit
* The toxicity from previous imatinib or other treatment has not been recovered ≤ grade 1 according to CTCAE 3.0
* Have surgery or radiotherapy within 4 weeks or have temporary radiotherapy for palliative treatment within 2 weeks
* A variety of factors that affect the oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction)
* Other cancer diagnosed within past 5 years or currently suffering , but other than cure basal cell carcinoma and cervical carcinoma in situ
* Within 12 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc
* Uncontrollable thyroid dysfunction, even using medical therapy
* Preexisting arrhythmia (including QT interval ≥ 450ms for male and 470ms for female) and ≥ grade I heart failure
* Patients with uncontrollable hypertension after using single agent therapy (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg).
* Known acute or chronic active hepatitis
* Immunodeficiency: HIV positive, or other acquired immunodeficiency, congenital immunodeficiency, or organ transplantation
* Less than 4 weeks from the last clinical trial
* Child bearing or pregnancy female. Potential child bearing female must have a negative urine or serum pregnancy test result before initiating.
* All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test drug.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.
* Mental disorders history, or Psychotropic drug abuse history
* Abuse of Psychiatric drugs or dysphrenia
* Other reasons from investigators' judgement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 12 weeks

SECONDARY OUTCOMES:
Objective Response Rate | 12 weeks
Progression free survival | 24 months
Overall survival | 96 months
Incidence of adverse events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Bayi Hospital, Nanjing, Jiangsu, China